CLINICAL TRIAL: NCT02612792
Title: Platelet Rich Fibrin Combined With 1.2% Atorvastatin Gel in Treatment of Mandibular Degree II Furcation Defects: a Randomized Controlled Clinical Trial
Brief Title: Platelet Rich Fibrin+1.2% Atorvastatin in Treatment of Mandibular Degree II Furcation Defects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and Head, Dept of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014U
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Furcation Defects
MeSH Terms: conditions — Furcation Defects | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Scaling and Root Planing (SRP) with Open flap debridement (OFD) alone for treating furcation defect
  Interventions: Procedure: Open flap debridement (OFD)
- Group 2 (Active Comparator): SRP with Open flap debridement (OFD) with Platelet rich fibrin (PRF) for treating furcation defect
  Interventions: Procedure: OFD with Platelet rich fibrin (PRF)
- Group 3 (Active Comparator): SRP with Open flap debridement (OFD) with Platelet rich fibrin (PRF)+1.2% Atorvastatin for treating furcation defect
  Interventions: Procedure: OFD with Platelet rich fibrin (PRF)+1.2% Atorvastatin (Drug) in gel form

INTERVENTIONS:
Procedure: Open flap debridement (OFD) — Open flap debridement (OFD) alone
  Arms: Group 1
Procedure: OFD with Platelet rich fibrin (PRF) — Open flap debridement (OFD) with Platelet rich fibrin (PRF) placement
  Arms: Group 2
Procedure: OFD with Platelet rich fibrin (PRF)+1.2% Atorvastatin (Drug) in gel form — Open flap debridement (OFD) with Platelet rich fibrin (PRF)+1.2% Atorvastatin gel placement
  Arms: Group 3

SUMMARY:
The present study was designed to explore the effectiveness of PRF combined with 1.2% ATV gel in treatment of mandibular degree II furcation defects in comparison to PRF and open flap debridement (OFD) alone.

DETAILED DESCRIPTION:
Background: A variety of regenerative materials have been tried since many years for the treatment of furcation defects. Platelet-rich fibrin (PRF), a pool reservoir of platelet concentrate with growth factors and Atorvastatin (ATV), a potent member of statin group are known to promote periodontal tissue regeneration. The aim of the present study is to explore the effectiveness of PRF combined with 1.2% ATV gel in treatment of mandibular degree II furcation defects in comparison to PRF and open flap debridement (OFD) alone.

Methods: Eighty two mandibular furcation defects were treated with either OFD alone (Group 1), OFD with PRF (Group 2), and OFD with PRF+1.2% ATV gel (Group 3).Clinical parameters like probing depth (PD), relative vertical clinical attachment level (RVCAL), relative horizontal clinical attachment level (RHCAL), modified sulcus bleeding index (mSBI) and site specific plaque index (PI) were recorded at baseline and 9 months post-operatively. The radiological assessment of bone defect fill was done at baseline and 9 months, using computer-aided software.

ELIGIBILITY:
Inclusion Criteria:

* Buccal degree II furcation defects in endodontically vital, asymptomatic mandibular first and second molars with a radiolucency in the furcation area on an intraoral periapical radiograph with probing depth (PD) ≥ 5mm and horizontal ≥ PD 3mm after phase I therapy i.e, scaling and root planing (SRP);
* No history of antibiotic or periodontal therapy in the preceding 6 months.

Exclusion Criteria:

* Aggressive periodontitis patients
* Systemic conditions known to affect the periodontal status;
* Medications known to affect the outcomes of periodontal therapy;
* Hematological disorders and insufficient platelet count (<100,000/mm3);
* Pregnancy/lactation;
* Smoking and tobacco use in any form
* Immunocompromised individuals;
* Those having unacceptable oral hygiene (plaque index [PI] >1.5).
* Teeth with furcation involvement, non-vital teeth, and carious teeth indicated for restorations and mobility of at least grade II were also excluded.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
. Radiographic bone fill assessed in percentage | baseline to 9 months
  assessed in percentage

SECONDARY OUTCOMES:
probing depth measured in mm | baseline to 9 months
  measured in mm
Relative vertical attachment level measured in mm | baseline to 9 months
  measured in mm
Relative horizontal attachment level measured in mm | baseline to 9 months
  measured in mm
modified sulcus bleeding index | baseline to 9 months
  0-3 scale
plaque index | baseline to 9 months
  0-3 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India